CLINICAL TRIAL: NCT05509478
Title: Lenvatinib Combined With PD-1 Inhibitors as First-line Treatment for Unresectable/Advanced Biliary Tract Carcinoma：a Multicenter,Single-arm,Phase II Study
Brief Title: Lenvatinib Combined With PD-1 Inhibitors as First-line Treatment for Unresectable/Advanced Biliary Tract Carcinoma
Acronym: LEADER-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstJlinU
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Cancer; PD-1 inhibitors; lenvatinib
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — lenvatinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib+PD-1 inhibitors (Experimental): Participants received lenvatinib capsules 8 mg , orally, once daily (QD) PD-1 inhibitors in this study include, but not limited to, Pembrolizumab, nivolumab, sintilimab, toripalimab, etc. The usage and dosage refer to label information or other clinical study
  Interventions: Drug: Lenvatinib; Drug: PD-1 inhibitors

INTERVENTIONS:
Drug: Lenvatinib — 8 mg once daily (QD) oral dosing.
  Other Names: E7080, Lenvima
Drug: PD-1 inhibitors — Regular dose intravenously every 3 weeks

SUMMARY:
This is a multi-center, single-arm,phase Ⅱ study to evaluate the efficacy and safety of Lenvatinib in combination with PD-1 inhibitors as first-line treatment in patients with unresectable advanced Biliary Tract Carcinoma (BTC)

ELIGIBILITY:
Inclusion Criteria:

1. Patients had good compliance, understood the study procedure, and signed written informed consent
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 2, Patients cannot tolerate chemotherapy or refuse to receive chemotherapy for any reason.
3. Pathologically or cytologically confirmed biliary tract cancer
4. Patients who are advanced and/or unresectable after imaging and multidisciplinary consultation
5. Patients must have at least one measurable lesion as defined by RECIST 1.1
6. Survival expectation of 12 weeks or longer after beginning of study treatment
7. The major organs meeting the following criteria:

   Adequate bone marrow function,defined as: Hemoglobin (HGB) ≥80g/L;Neutrophil absolute count (ANC) ≥1.0×10^9/L;Platelet (PLT) ≥60×10^9/L

   Adequate liver function, defined as: aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤ 2.5× upper limit of normal (ULN) ( ≤ 5.0 × ULN for participants with the liver transplantion);Serum total bilirubin（STB） <1.5×ULN

   Adequate renal function ，defined as：Serum creatinine was within 1.5 times the normal range
8. Patients requiring biliary stent implantation must complete the procedure at least 14 days before enrollment

Exclusion Criteria:

1. Allergy to Lenvatinib or PD-1 inhibitors
2. Patients who have had other malignancies within the past 2 years (except cured carcinoma in situ and basal cell carcinoma of the skin)
3. Patients who have previously received systemic therapy, except for permitted neoadjuvant/adjuvant therapy, neoadjuvant/adjuvant therapy should be completed at least 4 months before diagnosis of advanced and/or unresectable disease
4. Patients with ampullary carcinoma are excluded (patients with mixed HCC/ BTC may be considered)
5. Active autoimmune disease requiring systemic treatment (i.e. corticosteroids or immunosuppressive drugs) within the past 2 years.Alternative therapies (e.g., thyroxine, insulin, or physical corticosteroid replacement for adrenal or pituitary insufficiency) are not considered systemic and permitted
6. Major surgery prior to initiation of the study intervention and insufficient recovery from surgery and/or surgical complications
7. Radiation therapy was received within 2 weeks prior to initiation of study therapy. Or the subject must have recovered from all radiation-related toxicity, not required corticosteroids, and have not experienced radiation pneumonia; Palliative radiotherapy for non-central nervous system (CNS) disease (≤2 weeks) allows a washout period of 1 week (if deemed safe by the investigator)
8. Patients after organ transplantation
9. Known to have active tuberculosis (TB: tubercle bacilli)
10. Complete or incomplete intestinal obstruction
11. Have serious comorbidities that may affect study administration or evaluation of study results, such as HIV positive, active chronic HBV/HCV, clinically severe (i.e., active) heart disease, uncontrolled epilepsy, central nervous system disease, or psychiatric disorders;
12. Patients considered unsuitable for study judged by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 12-months
  ORR was assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. ORR was defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR). Confirmation of CR or PR was performed at least 28 days following the initial achievement of the response

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 12-months
  DCR was assessed by the investigator based on RECIST 1.1. DCR was defined as the percentage of participants whose BOR was CR, PR or SD
Progression-free Survival (PFS) | 12-months
  PFS was assessed by the investigator based on RECIST 1.1. PFS was defined as the time from the date of first dose to the date of last documentation of disease progression or date of death from any cause, whichever occurred first. For participants who did not have an event, PFS were censored. PFS was calculated using Kaplan-Meier method
Overall Survival (OS) | 24-months
  OS was defined as the time from the date of first dose to the date of death from any cause. For the participants who were alive or unknown, OS was censored on the last date participant was known to be event-free or date of data-cut-off. OS was calculated using the Kaplan-Meier method.
Overall Survival (OS) Rate at 9 months | 9-months
  OS was defined as the time from the date of first dose to the date of death from any cause. For the participants who were alive or unknown, OS was censored on the last date participant was known to be event-free or date of data-cut-off.
Overall Survival (OS) Rate at 12 months | 12-months
  OS was defined as the time from the date of first dose to the date of death from any cause. For the participants who were alive or unknown, OS was censored on the last date participant was known to be event-free or date of data-cut-off.

CONTACTS AND LOCATIONS:
Locations (1):
- Liu Bo, Changchun, Jilin, China